CLINICAL TRIAL: NCT00674999
Title: Project Title The Treatment of Partial Thickness Burns: Treated Amnion Versus Currently in Use Topical Medications
Brief Title: Use of Amnion on Partial Thickness Burns
Acronym: Amnion
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Hurricane- terminated study due to skin bank being destroyed
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 05-040
Record Dates: First submitted 2007-12-26; First posted 2008-05-08 (Estimated); Last update posted 2012-11-15 (Estimated); Status verified 2012-11

CONDITIONS: Burn
Keywords: Burn; Partial thickness burn
MeSH Terms: conditions — Burns | interventions — cancer procoagulant; bacitracin, polymyxin B drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): Amnion with processing procedures involving the use of trypsin-Edetic Acid(EDTA)
  Interventions: Biological: Amnion
- 2 (Experimental): Amnion with processing procedures involving the use of Dispase II
  Interventions: Biological: Amnion
- 3 (Active Comparator): Prepared Antibiotic ointment Polysporin, Bacitracin and Mycostatin
  Interventions: Drug: Polysporin/Bacitracin/Mycostatin

INTERVENTIONS:
Biological: Amnion — Application of Amnion with processing procedures involving the use of trypsin-EDTA
  Arms: 1
Biological: Amnion — Application of Amnion with processing procedures involving the use of Dispase II
  Arms: 2
Drug: Polysporin/Bacitracin/Mycostatin — Application of Prepared antibiotic ointment: Polysporin, Bacitracin and Mycostatin combined
  Arms: 3

SUMMARY:
To determine if Amnion, used on partial thickness burn injuries would provide an improvement in rate of healing, pain control and scarring as compared to standard medical treatments.

ELIGIBILITY:
Inclusion Criteria:

* Partial thickness burn injury.
* >2% burn injury.
* Ages 0-100 years.

Exclusion Criteria:

* Patients not expected to survive

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2005-06; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Length of time to 95% healing of treated burn wounds | Assessment daily until 95 % healed

SECONDARY OUTCOMES:
Length of hospital stay | Measured at hospital discharge
Incidence of infection | Measure daily until complete wound healing
Amount of daily pain until wound is healed with different treatments. | Daily until wound is completely healed.
Amount of scaring with different treatments | From injury to 2 years post burn

CONTACTS AND LOCATIONS:
Overall Officials: David N Herndon, MD, Principal Investigator — University of Texas